CLINICAL TRIAL: NCT01790217
Title: GERMAN TARCEVA NON-INTERVENTIONAL STUDY in 1st Line Treatment of NSCLC EGFR Mutation Positive Patients
Brief Title: An Observational Study of Tarceva (Erlotinib) in First Line in Patients With Advanced EGFR Mutation-Positive Non-Small Cell Lung Cancer (GERTAC)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML27895
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate the efficacy and safety of Tarceva (erlotinib) in first-line therapy in patients with locally advanced or metastatic EGFR mutation-positive non-small cell lung cancer. Eligible patients, for whom the treating physician has decided to initiate treatment with Tarceva according to the local label will be followed for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Locally advanced or metastatic EGFR mutation-positive non-small cell lung cancer
* Patients for whom the treating physician has decided to initiate first-line therapy with Tarceva in accordance with the Summary of Product Characteristics and local guidelines

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced or metastatic EGFR mutation positive non-small cell lung cancer
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2012-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Progression-free survival rate at 18 months | 3.5 years

SECONDARY OUTCOMES:
Response rate (complete response/partial response) by type of mutation | 3.5 years
Percentage of patients with remission | 3.5 years
Progression-free survival (overall/stratified) | 3.5 years
Overall survival (overall/stratified) | 3.5 years
Tolerability: Incidence of fatigue, rash, diarrhea | 3.5 years
Safety: Incidence of serious adverse events | 3.5 years
Dose modifications/withdrawals | 3.5 years
Symptom control (cough, dyspnea) | 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Oldenburg, Germany